CLINICAL TRIAL: NCT05061394
Title: Changes in Peak Fat Oxidation and Aerobic Fitness During Pre-season in Sub-elite Football Players
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: VentriJect ApS (Industry); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Professor, University of Copenhagen
Other Study IDs: VentriJect Football Study
Record Dates: First submitted 2021-03-10; First posted 2021-09-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Sub-elite Football Players
Keywords: Peak fat oxidation; Aerobic fitness; Football players; Treadmill running; Fatmax; Pre-season training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Second division football players: Players competing in the third best league in Denmark
- "Danmarkserien" football players: Players competing in the fourth best league in Denmark

SUMMARY:
Cross-sectional studies clearly demonstrate that the maximal fat oxidation (MFO, onwards referred to as peak fat oxidation, PFO) and the intensity at which it occurs (Fatmax) are higher in trained compared with untrained men and women (Maunder et al. 2018; Nordby et al. 2006; Lima-Silva et al. 2010). Furthermore, a recent study in endurance-trained males have shown a relationship between PFO and performance in an Ironman triathlon (Frandsen et al. 2017). The interest of PFO and Fatmax in endurance sports is centered on the speculation that increased fat oxidation rates during exercise would benefit endurance performance (> 4 hours) due to a glycogen sparing effect. Furthermore, it is speculated that the high amount of low-intensity training (70-80%), as seen with elite endurance athletes, might be essential in order to increase the fat oxidation capacity. However, when PFO is compared across an athletic population, football players have similar values as endurance-trained athletes (Randell et al. 2016; Randell et al. 2019; Frandsen et al. 2017), which is somewhat surprising when the different training regimes are considered.

It is noteworthy that the variations in PFO in various types of athletes and football players are considerable (Randell et al. 2016). However, different playing position in football has different work requirements, thus it might be that some of the variation seen in PFO could be related to the different playing position.

To our knowledge, no study has previously looked at the variations in fat oxidation capacity before and after a training period in athletes. Therefore, the aim of the present study is to investigate changes in peak fat oxidation and aerobic fitness during a pre-season training period in sub-elite football players. A secondary aim is to investigate if the changes are related to specific playing positions on the field. The overall hypothesis is that a pre-season training period would increase the fat oxidation capacity and aerobic fitness, and that the changes are related to specific player positions.

DETAILED DESCRIPTION:
Three sub-elite football teams in the Copenhagen area will be recruited for the study. The study will include two visits to our laboratory and field tests during the pre-season.

Before the participants volunteered to participate and signed a written informed consent form, the participants received both written and oral information about the content and possible risks associated with the study.

The participants arrived at the laboratory after an overnight fast (from latest 10pm). Furthermore, the participants were asked to avoid strenuous exercise 48 hours prior to the test day and eat a habitual diet, which had to be replicated before the second visit.

Testing at our laboratory includes:

* Measurements of height and weight anthropometry.
* Measurement of body composition using a Dual-energy X-ray absorptiometry (DXA) scan.
* Measurement of VO2max using a non-exercise testing method based on seismocardiography.
* Collection of a 15 ml resting venous blood sample for measurements of resting levels of hormones, metabolites and lipids in the blood plasma.
* Measurement of PFO and Fatmax during a graded submaximal running test on a motor driven treadmill.
* Measurement of VO2max on a motor driven treadmill.
* A questionnaire regarding previous and current football level, numbers of active years, playing position etc.

Procedure and analysis:

DXA scanning: The participants will be placed in the supine position in the DXA scanner (Lunar iDXA, GE Healthcare) after voiding and while wearing minimal clothing.

Blood samples: The blood samples will be collected from the vein cubiti medialis in the forearm. The blood will be sampled in iced BD vacutainers (5 mL Aprotinin, 4 mL EDTA and 2 mL Lithium Heparin) and immediately centrifuged at 4000 g for 10 minutes at 4⁰C (Rotina 380R, Hettich). The plasma will be collected and stored at -80⁰C for later analyzes of resting levels of metabolites, lipids and hormones.

The concentrations of hemoglobin, hematocrit, glucose and lactate will be immediately analyzed though sampling of 2 mL blood in a specialized syringe (safePICO Aspirator, Radiometer) and using an automatic analyzer (ABL800 Flex, Radiometer).

Exercise testing: The participants will perform a graded exercise test on a motor driven treadmill (Woodway Pro XL, Woodway USA Inc) with breath-by-breath measurements of pulmonary gas exchange by an automated online system (Quark CPET, Cosmed) throughout the test.

The protocol is adapted from Randell et al. 2019 with minor adjustments.

The protocol will start with a resting period with the participant sitting on a chair on the treadmill for 5 min. The exercise will hereafter commence at 6 km/h with a 1% incline for 5 minutes, where after the speed will be increased with 2 km/h every 3 minutes until the respiratory exchange ratio exceed 1.00. Subsequently, the incline will increase 2% every minutes until voluntary exhaustion, while the speed is held constant.

Participants will be wearing a chest strapped heart rate monitor (Garmin HRM-Tri, Garmin Forerunner 735XT, Garmin Ltd) with continuous heart rate measures during the test. Furthermore the participants, will be asked about perceived exhaustion on the 6-20 Borg scale directly following exhaustion.

The field tests will include three Yo-Yo intermittent Recovery level 2 test (YYIR2) and session-RPE (rate of perceived exertion (1-10 scale) for every training session. The YYIR2 will be scheduled with one in the second week of training, one midway and one during the last week of training before the start of the competitive season.

Statistical analysis:

All data will be checked for normal distribution (Shapiro-Wilk test) and equal variance (Brown- Forsythe test). The significant level is p<0.05.

Systematic differences in PFO, aerobic fitness, body composition and resting pre exercise blood values before and after the pre-season training period will be analyzed with a paired t test.

Pearson correlation analysis will be conducted with relevant resting pre exercise blood values and PFO, aerobic fitness and body composition in order to analyze association in possible differences between pre and post testing. Additionally, relevant resting pre exercise blood values will furthermore be analyzed with a coefficient of variation (CV%) analysis in order to look at the day-to-day variation.

In order to answer our secondary aim, a two-way ANOVA with repeated measures will be applied to analyze any effect of time and specific player position group in PFO and aerobic fitness. A post-hoc Sidak's multiple comparisons test will be applied when a significant effect of time or specific player positon group is found.

The project was approved by the Science Ethical commitee of the greater region of Copenhagen (H-20019103) the 3rd of July 2020. The protocol of the study adhered to the principles of the Helsinki declaration

ELIGIBILITY:
Inclusion Criteria:

* Sub-elite football player

Exclusion Criteria:

* Cardiovascular and/or metabolic disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sub-elite football players from three local football clubs in the Copenhagen region
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in Peak Fat Oxidation During Pre-season in Sub-elite Football Players | From January until April
  Peak Fat Oxidation (PFO) will be measured before and after pre-season in Sub-elite Football players, and pulmonary gas exchange will be measured during the treadmill running protocol as previously described. The fat oxidation rates will be calculated using the stoichiometric equations described by Frayn, with the assumption that urinary nitrogen excretion is negligible: Fat oxidation (g⋅min-1) = (1.67 ⋅ VȮ2) - (1.67 ⋅ V̇CO2). A 3nd-degree polynomial regression will be applied to determine PFO and the intensity at which it occurs (Fatmax) for each test individually. Changes in PFO from baseline and after 8 week pre-season will be measured and reported.
We will measure Aerobic Fitness before and after a Pre-season in Sub-elite Football Players | From January until April
  Aerobic Fitness will be measured before and pre-season in Sub-elite Football players, and pulmonary gas exchange measurements will be measured during the treadmill running protocol as previously described. VO2max will be reported both as an absolute value (ml/min) and relative to body-weight (ml/min/kg). The VO2max is determined as the highest value measured over consecutive 30 seconds. Changes in VO2max from baseline and after 8 week pre-season will be measured and reported.

SECONDARY OUTCOMES:
To investigate if the possible changes in Peak Fat Oxidation are related to specific playing positions on the field | From January until April
  The football players are divided into five different playing position (Goalkeeper, Center backs, Wingers, Midfielder, Striker) based on a questionnaire. The possible changes in the measured Peak Fat Oxidation from baseline to post pre-season will be compared between the different playing positions.
To investigate if the possible changes Aerobic Fitness are related to specific playing positions on the field | From January until April
  The football players are divided into five different playing position (Goalkeeper, Center backs, Wingers, Midfielder, Striker) based on a questionnaire. The possible changes in the measured Aerobic Fitness from baseline to post pre-season will be compared between the different playing positions.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, Professor, Principal Investigator — Department of Biomedical Sciences, Faculty of Health and Medical Sciences, University of Copenhagen
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randell RK, Carter JM, Jeukendrup AE, Lizarraga MA, Yanguas JI, Rollo I. Fat Oxidation Rates in Professional Soccer Players. Med Sci Sports Exerc. 2019 Aug;51(8):1677-1683. doi: 10.1249/MSS.0000000000001973. PMID 30845048
- [Background] Randell RK, Rollo I, Roberts TJ, Dalrymple KJ, Jeukendrup AE, Carter JM. Maximal Fat Oxidation Rates in an Athletic Population. Med Sci Sports Exerc. 2017 Jan;49(1):133-140. doi: 10.1249/MSS.0000000000001084. PMID 27580144
- [Background] Maunder E, Plews DJ, Kilding AE. Contextualising Maximal Fat Oxidation During Exercise: Determinants and Normative Values. Front Physiol. 2018 May 23;9:599. doi: 10.3389/fphys.2018.00599. eCollection 2018. PMID 29875697
- [Background] Nordby P, Saltin B, Helge JW. Whole-body fat oxidation determined by graded exercise and indirect calorimetry: a role for muscle oxidative capacity? Scand J Med Sci Sports. 2006 Jun;16(3):209-14. doi: 10.1111/j.1600-0838.2005.00480.x. PMID 16643200
- [Background] Lima-Silva AE, Bertuzzi RC, Pires FO, Gagliardi JF, Barros RV, Hammond J, Kiss MA. Relationship between training status and maximal fat oxidation rate. J Sports Sci Med. 2010 Mar 1;9(1):31-5. eCollection 2010. PMID 24149383
- [Background] Frandsen J, Vest SD, Larsen S, Dela F, Helge JW. Maximal Fat Oxidation is Related to Performance in an Ironman Triathlon. Int J Sports Med. 2017 Nov;38(13):975-982. doi: 10.1055/s-0043-117178. Epub 2017 Oct 19. PMID 29050040